CLINICAL TRIAL: NCT02089308
Title: Nicotine Patch - Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: V00116 TD 1 06; 2013-005290-47 (EudraCT Number)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Smokers
Keywords: Smoking cessation; Nicotine; Tobacco Use Disorder; Central Nervous System Agents
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

ARMS (2):
- Treatment-Sequence 1 (Other): Subjects will be randomly assigned to one of 2 treatment-sequence groups with 2 treament periods.
  Treatment -Sequence 1 : Period 1 (test drug) + period 2 (reference)
  The duration of each treatment period will be 3 days. Each patch will be applied for 24 hours.
  Interventions: Drug: Test treatment : V0116 transdermal patch; Drug: Reference treatment : Nicotine transdermal patch
- Treatment-Sequence 2 (Other): Subjects will be randomly assigned to one of 2 treatment-sequence groups with 2 treament periods.
  Treatment-sequence 2 : Period 1 (reference) + period 2 (test drug)
  The duration of each treatment period will be 3 days. Each patch will be applied for 24 hours.
  Interventions: Drug: Test treatment : V0116 transdermal patch; Drug: Reference treatment : Nicotine transdermal patch

INTERVENTIONS:
Drug: Test treatment : V0116 transdermal patch
Drug: Reference treatment : Nicotine transdermal patch

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a new transdermal nicotine patch to that of a reference formulation following repeated applications

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject aged 18 to 45 years (inclusive)
* Current Smoker of >or = 5 and < or = to 15 cigarettes/day
* Fagerström score < or =5 at selection
* Absence of any clinically significant abnormal findings at physical examination, vital sign, Electrocardiogram ECG, biological examinations in the investigator's opinion.

Exclusion Criteria:

* Presence of any significant medical findings or significant history (in particular any cardio-vascular disease, severe renal or hepatic insufficiency, current gastric or duodenal ulcer) that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator
* Any visible skin disorder, abnormal skin pigmentation or dermatologic disease liable to interfere with use or safety assessment of a transdermal patch

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | During the third application of each period,12 time points up to 24h after the application
Time to Maximum Concentration (Tmax) | During the third application of each period,12 time points up to 24h after the application
Area under the plasma concentration-time curve (AUC) | During the third application of each period, 12 time points up to 24h after the application

CONTACTS AND LOCATIONS:
Locations (1):
- Gières, France